CLINICAL TRIAL: NCT05140967
Title: Effects of Endurance Training Intensity on Exercise Capacity, Body Composition, and Appetite Regulation in Cystic Fibrosis
Brief Title: Effects of Training Intensity on Physical Fitness and Body Composition in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kiel (Other)
Collaborators: Fachklinik Satteldüne der DRV Nord (Unknown); University of Kiel, Arbeitsbereich Sportmedizin und Trainingswissenschaften (Unknown); Strandklinik St. Peter-Ording (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Anja Bosy-Westphal, Prof. Dr. Dr. Anja Bosy-Westphal, University of Kiel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABW-2021-CF
Record Dates: First submitted 2021-10-29; First posted 2021-12-02 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Cystic Fibrosis
Keywords: Exercise training; High Intensity Interval Training (HIIT); Moderate Intensity Continuous Training (MICT); Exercise capacity; Peak Oxygen uptake (VO2peak); Body-composition; Subjective appetite and satiety ratings; Appetite regulating hormones; Health related quality of life; Habitual physical activity; ad libitum energy intake
MeSH Terms: conditions — Cystic Fibrosis | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Intensity Interval Training (A) (Experimental): Exercise training with intermittent bouts of high intensity
  Interventions: Other: High Intensity Interval Training (HIIT)
- Moderate Intensity Continous Training (B) (Experimental): Exercise training with constant workload
  Interventions: Other: Moderate Continuous Intensity Training (MICT)

INTERVENTIONS:
Other: High Intensity Interval Training (HIIT) — High Intensity Interval Training
  Arms: High Intensity Interval Training (A)
Other: Moderate Continuous Intensity Training (MICT) — Moderate Intensity Continuous Training
  Arms: Moderate Intensity Continous Training (B)

SUMMARY:
Aim of the randomized controlled trial is to investigate the effects of endurance training with different intensities on physical performance, body composition and appetite regulation in people with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of cystic fibrosis by at least 2 sweat tests and / or by the presence of two CF mutations,
* willingness to participate in and to comply with the research project procedure,
* written informed consent of patients,
* age ≥ 18 years,
* FEV1 of pred. ≥ 40%,
* Stable condition (as indicated by absence of one or more signs: new or increased haemoptysis, increased malaise, fatigue or lethargy, temperature over 38°C, weight loss, sinus pain and a decrease in pulmonary function by 10% or more)

Exclusion Criteria:

* Severe pulmonary exacerbation,
* cor pulmonale,
* musculoskeletal discomfort that makes a regular exercise training impossible,
* untreated CF-related diabetes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
change in Peak Oxygen Uptake | at baseline and after 4 weeks of exercise training program
  measured with peak Oxygen uptake (VO2) in percent predicted
change in Peak Workload | at baseline and after 4 weeks of exercise training program
  measured with peak Workload in percent predicted
change body fat mass index | at baseline and after 4 weeks of exercise training program
  measured with body fat mass index (FMI) in kg / m*2
change in Body fat free mass index | at baseline and after 4 weeks of exercise training program
  measured with fat free body mass index (FFMI) in kg / m*2

SECONDARY OUTCOMES:
change in Forced Expiratory Volume in 1 second | at baseline and after 4 weeks of exercise training program
  measured with Forced Expiratory Volume in 1 second (FEV1) in percent predicted
change in Health related quality of life | at baseline and six and twelve months after completion of exercise training program
  measured with the Cystic Fibrosis Questionnaire Revised (CFQ-R); 9 Quality of life domains: Physical, role/school, vitality, emotion, social, body image, eating, treatment burden, health perceptions: 3 symptom scales: Weight, respiratory, and digestion Scores range from 0 to 100, with higher scores indicating better health.
appetite control - subjective feeling of hunger | at baseline and after 4 weeks of exercise training program
  measured with visual analogue scales. The scale consists of a 10 cm vertical line anchored with "not hungry at all" at the left side and with "extremely hungry" at the right side.

CONTACTS AND LOCATIONS:
Overall Officials: Anja Bosy-Westhphal, Prof, PhD, MD, Study Chair — Insitute of Human Nutrition, University of Kiel
Locations (2):
- Germany (2):
  - Fachklink Satteldüne der DRV Nord, Nebel / Amrum, Schleswig-Holstein
  - Strandklinik St. Peter-Ording, Sankt Peter-Ording, Schleswig-Holstein